CLINICAL TRIAL: NCT00976677
Title: Randomized Double-Blind Placebo Controlled Phase II Trial Evaluating Erlotinib in Non-Smoking Patients With (Bevacizumab-Eligible and Ineligible) Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Carboplatin, Paclitaxel, and Bevacizumab With or Without Erlotinib Hydrochloride in Treating Non-Smokers With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2011-01967; NCI-2011-01967 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E2508; CDR0000654212; E2508 (Other: Eastern Cooperative Oncology Group); E2508 (Other: CTEP); U10CA021115 (NIH)
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2013-07-22 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2013-12

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Paclitaxel; Taxes; Carboplatin; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (Active Comparator): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes (with or without bevacizumab IV over 30-90 minutes) on day 1. Patients also receive placebo PO QD on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients with stable or responding disease may continue to receive placebo (with or without bevacizumab) as above in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel; Drug: carboplatin; Biological: bevacizumab
- Arm II (Experimental): Patients receive paclitaxel and carboplatin (with or without bevacizumab) as in arm I. Patients also receive erlotinib hydrochloride PO QD on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients with stable or responding disease may continue to receive erlotinib hydrochloride (with or without bevacizumab) as above in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: paclitaxel; Drug: carboplatin; Biological: bevacizumab

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
  Arms: Arm II
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF

SUMMARY:
This randomized phase II trial studies how well carboplatin, paclitaxel, and bevacizumab work with or without erlotinib hydrochloride in treating non-smokers with advanced non-small cell lung cancer. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether giving combination chemotherapy together with bevacizumab is more effective with or without erlotinib hydrochloride in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression-free survival (PFS) of non-smokers with advanced non-small cell lung cancer (NSCLC) randomized to standard of care (either carboplatin/paclitaxel with or without bevacizumab), or standard of care plus erlotinib hydrochloride.

SECONDARY OBJECTIVES:

I. To evaluate the overall survival from day of randomization. II. To evaluate response rate. III. To evaluate relative toxicity. IV. To determine the frequency of epidermal growth factor receptor (EGFR) and Kras mutations in non-smokers with NSCLC and correlate mutation status with response rate and progression free survival.

V. To obtain blood and tissue specimens for further marker-based exploratory analyses regarding EGFR inhibitors.

VI. To evaluate EGFR positivity by fluorescence in situ hybridization (FISH) as a predictor of improved PFS in patients treated with erlotinib hydrochloride.

OUTLINE: This is a multicenter study. Patients are stratified according to gender and eligibility for bevacizumab therapy (ineligible vs eligible and willing to receive bevacizumab vs eligible and not willing to receive bevacizumab). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes (with or without bevacizumab IV over 30-90 minutes) on day 1. Patients also receive placebo orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients with stable or responding disease may continue to receive placebo (with or without bevacizumab) as above in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive paclitaxel and carboplatin (with or without bevacizumab) as in arm I. Patients also receive erlotinib hydrochloride PO QD on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients with stable or responding disease may continue to receive erlotinib hydrochloride (with or without bevacizumab) as above in the absence of disease progression or unacceptable toxicity.

Blood and tissue samples are collected for correlative laboratory studies.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease as defined by Response Criteria In Solid Tumors (RECIST) criteria
* Baseline measurements and evaluations of all sites of disease must be obtained =< 4 weeks (28 days) prior to randomization
* Eastern Cooperative Oncology Group (ECOG) performance status between 0-1
* No prior chemotherapy for lung cancer; prior chemotherapy for an unrelated condition is allowed if completed > 3 years prior to date of randomization
* Histological or cytologic evidence of non-small cell lung cancer
* Patients must not have any additional active, invasive malignancies requiring therapy
* Patients must have smoked less than or equal to 100 cigarettes in their lifetime
* Stage IV or IIIB (with pleural or pericardial effusion or multifocal pleural involvement) or recurrence after prior curative resection or definitive radiation
* Prior radiation therapy (RT) is allowed, provided RT has ended at least 2 weeks (14 days) prior to date of randomization; patients must have recovered from any adverse events related to the RT (except alopecia and grade 1 neuropathy); no previous irradiation to the only site of measurable disease, unless that site has had subsequent evidence of pathologic or radiologic progression
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin =< 1.5 mg/dl
* Creatinine =< 2.0 mg/dl
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvate transaminase (SGPT) =< 3 X institutional upper limit of normal (ULN)
* Women must not be pregnant or breast-feeding due to unknown interaction between erlotinib and the developing fetus or newborns potentially exposed to erlotinib by ingestion of lactated milk; all females of childbearing potential must have a blood test within 2 weeks prior to randomization to rule out pregnancy
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception
* Patients must not have clinically significant ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient must meet the following criteria:

  * Non-squamous histology
  * No antecedent hemoptysis
  * International normalized ratio (INR) =< 3 within 4 weeks (28 days) prior to randomization
* Patients may be on a stable regimen of therapeutic anticoagulation or may be receiving prophylactic anticoagulation of venous access devices, provided that coagulation studies met entry criteria; caution must be exercised for patients requiring anticoagulation, including treatment with low dose heparin or low molecular weight heparin for deep vein thrombosis (DVT) prophylaxis while on study due to an increased risk of bleeding with bevacizumab
* No history of untreated brain metastases NOTE: Recent data (PASSPORT, ATLAS, AIRES) suggest that bevacizumab can be given in patients with treated brain metastases; investigators can use their discretion in deciding whether to use bevacizumab in patients who fulfill these criteria
* Urine dipstick must be =< 0-1+ within 4 weeks (28 days) of randomization. If urine dipstick is > 1+ then the Urine Protein Creatinine (UPC) ratio must be calculated
* Patients must have no history of thrombotic or hemorrhagic disorders
* Patients with history of hypertension must be well-controlled (blood pressure [BP] =< 150/90 within 4 weeks [28 days] of randomization) and on a stable regimen of anti-hypertensive therapy (within 4 weeks of randomization)
* Patients must not have serious non-healing wound ulcer, bone fracture, or major surgical procedure within 28 days prior to randomization
* Patients with a known history of myocardial infarction or other evidence of arterial thrombotic disease (angina) will be allowed on study only if they have had no evidence of active disease for at least 6 months prior to randomization
* Patients must not have a history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to randomization
* Patients must not have significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomization
* Patients must not have clinically significant cardiovascular disease including:

  * History of cerebral vascular accident (CVA) within 6 months
  * New York Heart Association grade II or greater congestive heart failure
  * Serious and inadequately controlled cardiac arrhythmia
  * Clinically significant peripheral vascular disease (symptomatic with intermittent claudications or < 6 months from a bypass operation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Langer, Principal Investigator — Eastern Cooperative Oncology Group
Locations (108):
- United States (108):
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Saint Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - McFarland Clinic, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - UHHS-Chagrin Highlands Medical Center, Orange, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - Parkland Memorial Hospital, Dallas, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - Saint Paul Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to accrual on January 27, 2010 and was terminated on May 13, 2011 due to slow accrual. Final accrual was 10 patients.
Groups:
- Arm A: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes (with or without bevacizumab IV over 30-90 minutes) on day 1. Patients also receive an oral placebo once daily on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients with stable or responding disease may continue to receive placebo (with or without bevacizumab) as above in the absence of disease progression or unacceptable toxicity.
- Arm B: Patients receive paclitaxel and carboplatin (with or without bevacizumab) as in arm A. Patients also receive oral erlotinib hydrochloride once daily on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients with stable or responding disease may continue to receive erlotinib hydrochloride (with or without bevacizumab) as above in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 5 | 5
Completed | 0 | 0
Not Completed | 5 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Disease progression | 1 | 1
Not completed — Trial unblinded | 2 | 2
Not completed — Unknown/Missing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Median (Full Range); unit: years] | 53 [38 to 76] | 63 [60 to 75] | 62 [38 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined to be the time from randomization to progression of disease or death, whichever occurs first. Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Every 6 weeks during treatment and every 3 months in follow-up until disease progression or up to 5 years
Population: All eligible and treated patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 5 | 5
Months | 4.5 [4.5 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 15.5 [6.74 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Assessed every 21 days while on treatment and for 30 days after the end of treatment.
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 1/5 | 3/5
Other Adverse Events (participants affected / at risk) | 2/5 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=5) | Arm B (N=5)
Fatigue (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=5) | Arm B (N=5)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Fatigue (General disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Blurred vision (Eye disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less